CLINICAL TRIAL: NCT06203743
Title: Evaluation of Caudal Block and Ilioinguinal-ilioohypogastric Nerve Block Efficacy with Perfusion Index (PI) in Pediatric Inguinal Hernia Operations Under General Anesthesia
Brief Title: Evaluation of Caudal Block and Ilioinguinal-ilioohypogastric Nerve Block Efficacy with Perfusion Index (PI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Aycan KURTARANGİL DOĞAN, Doctor of anesthesiology and reanimation, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BYIEAH-AKD-01
Record Dates: First submitted 2023-12-11; First posted 2024-01-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Perfusion Index; Plethysmography; Anesthesia, Caudal; Nerve Block; Anesthesia, Regional; Child; Inguinal Hernia Unilateral
Keywords: Perfusion Index; plethysmography variability index; caudal block; ilioinguinal iliohypogastric nerve block; nerve block; Inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: The research is a prospective controlled, randomized, double-blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study randomization will be done in sealed envelopes using computer-generated randomization codes by a doctor who will not participate in patient follow-up. For the quality and standardization of the block with bupivacain, the caudal and ilioinguinal-iliohypogastric block will be performed by an anesthetist experienced in regional anesthesia. Postoperative Flacc pain scale, type and amount of additional analgesic will be recorded by a doctor blinded to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (No Intervention): Patients in this group will not undergo any block after LMA. PI, PVI, pulse, saturation, noninvasive arterial pressure values will be recorded before induction, after induction, after LMA, at 0, 5, 10, 15, 20, 25 and 30 minutes after the surgical incision and at the end of anesthesia. PI, PVI will be monitored with Radical-97TM Pulse CO-OximeterTM (Masimo Corp, Irvine, CA, USA) probe.
- caudal block group (Active Comparator): Patients in this group will receive a caudal block in the lateral decubitus position after LMA with 0.25% Buvasin® 0.5ml/kg. PI, PVI, pulse, saturation, noninvasive arterial pressure values before induction, after induction, after LMA, before applied block, after applied block (after surgical incision) 0., 5., 10., 15., 20., 25. It will be recorded at the 30th and 30th minutes and at the end of anesthesia. PI, PVI will be monitored with Radical-97TM Pulse CO-OximeterTM (Masimo Corp, Irvine, CA, USA) probe.
  Interventions: Procedure: caudal block group
- ilioinguinal-iliohypogastric nerve block group (Active Comparator): Patients in this group will undergo an ilioinguinal-iliohypogastric nerve block in the supine position under ultrasound guidance after LMA with 0.25% Buvasin® 0.5ml/kg. PI, PVI, pulse, saturation, noninvasive arterial pressure values before induction, after induction, after LMA, before applied block, after applied block (after surgical incision) 0., 5., 10., 15., 20., 25. It will be recorded at the 30th and 30th minutes and at the end of anesthesia. PI, PVI will be monitored with Radical-97TM Pulse CO-OximeterTM (Masimo Corp, Irvine, CA, USA) probe.
  Interventions: Procedure: ilioinguinal-iliohypogastric nerve block group

INTERVENTIONS:
Procedure: caudal block group — PI, PVI measurements and hemodynamic data will be compared between groups
  Arms: caudal block group
Procedure: ilioinguinal-iliohypogastric nerve block group — PI, PVI measurements and hemodynamic data will be compared between groups
  Arms: ilioinguinal-iliohypogastric nerve block group

SUMMARY:
The study is a prospective, randomised, controlled double-blind clinical trial. The primary aim was to evaluate the efficacy of caudal block and ilioinguinal-iliohypogastric nerve block with PI and PVI in pediatric inguinal hernia operations under general anesthesia. The secondary aim is to evaluate postoperative analgesic agent consumption and to evaluate the correlation of PI and PVI values with hemodynamic parameters. Pediatric patients between the ages of 2-8 years who are planned to undergo elective inguinal hernia operation will be included in the study. After the patients scheduled for inguinal hernia surgery are admitted to the operating room, routine monitoring will be performed as performed. In addition to routine monitoring, a Radical-97TM Pulse CO-OximeterTM (Masimo Corp, Irvine, CA, USA) probe will be attached to the toe to monitor PI and PVI. Patients will be given anaesthetic drugs as routinely administered. After LMA by randomisation by closed envelope method, caudal or ilioinguinal-iliohypogastric nerve block will be performed by an experienced anaesthetist as the investigators routinely perform in patients other than the control group.. PI, PVI, pulse, saturation, noninvasive arterial pressure values will be recorded before induction, after induction, after LMA, before applied block, after applied block (after surgical incision) at 0, 5, 10, 15, 20, 25 and 30 minutes and at the end of anaesthesia. All patients will be given paracetamol 10mg/kg iv, which is a routine intravenous (iv) analgesic, at the end of surgery. In case of perioperative complications, the complications will be recorded.

Flacc pain scale (Face, Legs, Activity, Cry, Consolability) will be applied at 0, 2, 6 hours postoperatively. Postoperative analgesic use and discharge time will be recorded. Flacc pain scale will be performed by an anaesthetist blinded to the study.

DETAILED DESCRIPTION:
The study is a prospective, randomised, controlled double-blind clinical trial. The primary aim was to evaluate the efficacy of caudal block and ilioinguinal-iliohypogastric nerve block with PI and PVI in pediatric inguinal hernia operations under general anesthesia. The secondary aim is to evaluate postoperative analgesic agent consumption and to evaluate the correlation of PI and PVI values with hemodynamic parameters. Pediatric patients between the ages of 2-8 years who are planned to undergo elective inguinal hernia operation will be included in the study.

ASA III-IV patients, patients with peripheral vascular disease, patients with diabetes mellitus, patients with neuromuscular disease, patients with bleeding disorders, patients with infection at the site of the block, patients with infection at the site of perfusion index probe adhesion, patients with bilateral inguinal hernia operation, patients with inguinal hernia operation with circumcision, patients with emergency operation, patients with mental retardation, patients who do not speak Turkish, patients with local anesthetic allergy, patients who do not give consent to participate in the study will not be included.

After the patients scheduled for inguinal hernia surgery are admitted to the operating room, routine monitoring will be performed as performed in the clinic. In addition to routine monitoring, a Radical-97TM Pulse CO-OximeterTM (Masimo Corp, Irvine, CA, USA) probe will be attached to the toe to monitor PI and PVI and covered with gauze to prevent exposure to ambient light. Patients will be given anaesthetic drugs as routinely administered (propofol 1-3mg/kg, fentanyl 1-2mcg/kg), followed by placement of an appropriately sized supraglottic airway device (LMA) and maintenance of anaesthesia with oxygen, air and sevoflurane. After LMA by randomisation by closed envelope method, caudal or ilioinguinal-iliohypogastric nerve block will be performed by an experienced anaesthetist as the investigators routinely perform in patients other than the control group. Caudal block is performed in the left lateral decubitus position after sterile conditions are provided, the sacral cornuas are palpated and a 25 gauge caudal needle (egemen international brand 25g 30 mm) is advanced at an angle of 45 degrees. After the needle hits the sacrum, the angle is reduced by retreating a few millimetres and the epidural area is reached in the sacral canal. After controlling the absence of blood and cerebrospinal fluid by negative aspiration, Buvasin® will be administered at a dose of 0.25%, 0.5 ml/kg. Ilioinguinal-iliohypogastric nerve block will be performed by placing the linear probe transversely-obliquely in the direction of the line connecting the spina iliaca anterior superior and the umbilicus under ultrasound guidance after sterile conditions are provided while the patient is in the supine position. The block needle (braun brand stimplex ultra 360 block needle) is inserted with in-plane technique in the same plane with the ultrasound probe. External and Internal Oblique Muscle and Transversus Abdominus Muscle layers and nerves are determined, needle tip localisation is determined, aspirated at frequent intervals and 0.25% Buvasin® 0.5ml/kg is given to the neurofascial plan. PI, PVI, pulse, saturation, noninvasive arterial pressure values will be recorded before induction, after induction, after LMA, before applied block, after applied block (after surgical incision) at 0, 5, 10, 15, 20, 25 and 30 minutes and at the end of anaesthesia. All patients will be given paracetamol 10mg/kg iv, which is a routine intravenous (iv) analgesic, at the end of surgery. In case of perioperative complications, the complications will be recorded.

Flacc pain scale (Face, Legs, Activity, Cry, Consolability) will be applied at 0, 2, 6 hours postoperatively. Postoperative analgesic use and discharge time will be recorded. Flacc pain scale will be performed by an anaesthetist blinded to the study.

ELIGIBILITY:
Inclusion Criteria:

* 2-8 years old
* Elective Inguinal hernia operation
* ASA I-II patients

Exclusion Criteria:

* <2 years to be >8 years old
* ASA III-IV patients
* Peripheral vascular disease
* Diabetes Mellitus patient
* Neuromuscular disease
* Bleeding disorder
* Infection in the area to be blocked
* Infection at the perfusion index probe adhesion site
* Bilateral inguinal hernia operation
* Inguinal hernia operation with circumcision
* Cases taken to emergency operation
* Mental retardation
* Not knowing Turkish
* Allergy to local anesthetics
* Refusal to participate in the research

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
PI and PVI | during the operation
  PI and PVI will be measured using a Radical-97TM Pulse CO-OximeterTM (Masimo Corp, Irvine, CA, USA) probe. PI, PVI and hemodynamic data will be used to evaluate the efficacy of the blocks and the pain status of the patients.

SECONDARY OUTCOMES:
FLACC pain scale | up to six hour
  Face, Legs, Activity, Cry, Consolability (FLACC) pain scale to be administered in the first 6 hours after surgery
Analgesic use | 1 day
  Amount and number of analgesics used postoperatively
Duration of discharge | 1 day
  Discharge time after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aycan Kurtarangil Doğan, Principal Investigator — akurtarangil@gmail.com
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No